CLINICAL TRIAL: NCT03019705
Title: An Examination of the Effects of Health-related Internet Use in Individuals With Pathological Health Anxiety Using Ambulatory Assessment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Principal Investigator, Sandra K. Hamann, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: C2-aA
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Health Anxiety
Keywords: Cyberchondria; health-related internet use; pathological health anxiety; ambulatory assessment
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants: Individuals with pathological health anxiety
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
The purpose of the current explorative study is to examine the effects of health-related internet use in individuals with pathological health anxiety using ambulatory assessment. In a naturalistic setting participants answer over a seven-day period questionnaires about their health-related internet use and its effects on affect, health anxiety and symptom severity in their usual daily lives.

DETAILED DESCRIPTION:
The internet is a popular method for obtaining information. Increasingly, it is also used to answer medical and health questions, because compared to other methods (e.g. going to the library or visiting a doctor) it has a number of advantages to offer like low costs, availability, easy accessibility, anonymity, and great diversity of information types and sources. 60 to 80 percent of internet users search online for medical information. In this context the term "cyberchondria" was coined in the media to describe the potentially detrimental effects of this behavior. The first studies in this field using self-report retrospective data showed that individuals with elevated levels of health anxiety seem to make increased use of the internet for this purpose and it seems to maintain health anxiety in the long-term. However, up until today little is known about the consequences of this behavior and the maintaining mechanism.

This observational study aims to investigate the effects of health-related internet use in individuals with pathological health anxiety in a naturalistic setting using ambulatory assessment. The variables of interest are monitored using time- and event-based sampling methods. Therefore, over a seven-day period participants answer seven times a day questionnaires on a mobile phone in their usual daily lives and additionally track the variables of interest in the moment the target behavior (health-related internet use) occurs. To our knowledge, this is the first study to investigate these relations using ambulatory assessment and therefore additionally aims to investigate the feasibility of this study design in this specific field of research.

ELIGIBILITY:
Inclusion Criteria:

* Pathological health anxiety according to the criteria of Fink et al., 2004
* Informed consent
* Sufficient German language skills
* Sufficient skills using a computer, a mobile phone and the internet

Exclusion Criteria:

* Suicidal tendency
* Clinical diagnosis of alcohol or drug abuse, acute schizophrenia
* Organic brain disorders
* Impairment of intelligence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: individuals with pathological health anxiety
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change of health anxiety before and after health-related internet use | Time-based sampling: every day at 9am, 11am, 1pm, 3pm, 5pm, 7pm and 9pm during seven days
  Self-created item. The occurence of health-related internet use is indicated by answering a question (yes/no) for a specific time period (e.g. between 9am and 11am), then the difference score for levels of health anxiety between these two time points is calculated.
Change of positive and negative affect before and after health-related internet use | Time-based sampling: every day at 9am, 11am, 1pm, 3pm, 5pm, 7pm and 9pm during seven days
  Short-form of the Positive Affect Negative Affect Schedule -State (PANAS-State) by Thompson (2007), translated into German.
  The occurence of health-related internet use is indicated by answering a question (yes/no) for a specific time period (e.g. between 9am and 11am), then the difference score for levels of health anxiety between these two time points is calculated.
Change of symptom severity before and after health-related internet | Time-based sampling: every day at 9am, 11am, 1pm, 3pm, 5pm, 7pm and 9pm during seven days
  Self-created item. The occurence of health-related internet use is indicated by answering a question (yes/no) for a specific time period (e.g. between 9am and 11am), then the difference score for levels of health anxiety between these two time points is calculated.
Change of health anxiety before and after health-related internet use | Event-based sampling: before and after every health-related internet use that is conducted during a seven-day-period
  Self-created item. Start and end of health-related internet use is indicated by the push of a special button on the mobile phone and triggers the presentation of this item.
Change of positive and negative affect before and after health-related internet use | Event-based sampling: before and after every health-related internet use that is conducted during a seven-day-period
  Short-form of the Positive Affect Negative Affect Schedule -State (PANAS-State) by Thompson (2007), translated into German.
  Start and end of health-related internet use is indicated by the push of a special button on the mobile phone and triggers the presentation of this questionnaire.
Change of symptom severity before and after health-related internet | Event-based sampling: before and after every health-related internet use that is conducted during a seven-day-period
  Self-created item. Start and end of health-related internet use is indicated by the push of a special button on the mobile phone and triggers the presentation of this item.

SECONDARY OUTCOMES:
frequency of occurence of health-related internet use | during seven days
  start of health-related internet use is recorded by the push of a special button on the mobile phone

CONTACTS AND LOCATIONS:
Overall Officials: Michael Witthoeft, Professor, Study Chair — Department of Clinical Psychology, Psychotherapy and Experimental Psychopathology, Johannes Gutenberg University Mainz